CLINICAL TRIAL: NCT01480440
Title: Prospective Post Market Clinical Follow-up Study of the Zimmer Trabecular Metal Reverse Should System Used in Primary or Revision Reverse Total Shoulder Arthroplasty
Brief Title: Outcomes Study of the Trabecular Metal (TM) Reverse Shoulder System
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMU2010-28E
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post-traumatic Arthritis; Ununited Humeral Head Fracture; Irreducible 3-and 4-part Proximal Humeral Fractures; Avascular Necrosis; Gross Rotator Cuff Deficiency; Revision Total Shoulder Arthroplasty
Keywords: Reverse Total Shoulder Arthroplasty (TSA); Reverse TSA; Osteoarthritis; Rheumatoid Arthritis; Post-traumatic arthritis; Ununited humeral head fracture; Irreducible 3-and 4-part proximal humeral fractures; Avascular necrosis; Gross rotator cuff deficiency; Failed total shoulder arthroplasty; Revision total shoulder arthroplasty
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Trabecular Metal Reverse Shoulder System: Patients requiring primary or revision reverse total shoulder arthroplasty who receive the Trabecular Metal Reverse Shoulder System
  Interventions: Device: Trabecular Metal Reverse Shoulder System

INTERVENTIONS:
Device: Trabecular Metal Reverse Shoulder System — Trabecular Metal Reverse Shoulder System used in primary or revision total shoulder arthroplasty
  Other Names: TM Reverse Shoulder System; TM Reverse System; TM Reverse

SUMMARY:
The objectives of this study are to obtain survival and outcome data on the Trabecular Metal Reverse Shoulder System when used in primary or revision reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
The objectives of this study are to obtain survival and outcome data on the Trabecular Metal Reverse Shoulder System when used in primary or revision reverse total shoulder arthroplasty. This will be done by analysis of standard scoring systems, radiographs and adverse event records. Data will be collected and analyzed to monitor pain, function, and survivorship and to confirm the performance of the Trabecular Metal Reverse Shoulder System.

Performance will be evaluated by monitoring the frequency and incidence of adverse events as well as by assessment of the overall pain and functional performances, survivorship, health status and radiographic parameters of all enrolled study subjects who receive the Trabecular metal Reverse Shoulder System.

Pain and functional performance will be measured using the American Shoulder and Elbow Surgeons (ASES) Shoulder Assessment and the Single Assessment Numeric Evaluation (SANE), survivorship will be based on removal or intended removal of the device, health status will be determined by evaluation of the Short Form Survey12 (SF-12) as well as Adverse Events (AEs) and radiographic parameters analysis of x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years of age;
* Patient is skeletally mature;
* Patient qualifies for primary or revision unilateral or bilateral reverse total shoulder arthroplasty based on physical exam and medical history including the following: osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, ununited humeral head fracture, irreducible 3-and 4-part proximal humeral fractures, avascular necrosis, gross rotator cuff deficiency or failed total shoulder arthroplasty (both glenoid and humeral components require revision);
* Patient is willing and able to provide written informed consent;
* Patient is willing and able to cooperate in the required post-operative therapy;
* Patient is willing and able to complete scheduled follow-up evaluations/questionnaires as described in the Informed Consent;
* Patient has participated in the Informed Consent process and has signed the Institutional Review Board (IRB)/Ethical Review Board (ERB) approved informed consent.

Exclusion Criteria:

* The patient is a prisoner;
* The patient is mentally incompetent or unable to understand what participation in the study entails;
* The patient is a known alcohol or drug abuser;
* The patient is anticipated to be non-compliant;
* The patient has one of the following compromising the affected limb: a significant injury to the upper brachial plexus, paralysis of the axillary nerve or a neuromuscular disease compromising the affected limb which would render the procedure unjustifiable;
* The patient has a local/systemic infection;
* The patient is known to be pregnant;
* The patient has marked bone loss;
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials;
* The patient is unwilling or unable to give consent or to comply with the follow-up program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each investigator will screen from his/her patients who suffer from osteoarthritis, rheumatoid arthritis, post-traumatic arthritis, ununited humeral head fracture, irreduciable 3-and 4-part proximal humeral fractures, avascular necrosis, gross rotator cuff dificiency or failed total shoulder arthroplasty (both glenoid and humeral components require revision) who meet the inclusion/exclusion criteria stated in the protocol
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 Years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Pain and Functional Performance | 10 Years
  Measurements will be based on the American Shoulder and Elbow Surgeons (ASES) Shoulder Assessment and the Single Assessment Numeric Evaluation (SANE)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Norton Orthopaedic & Sports Medicine, Louisville, Kentucky
  - The Rothman Institute, Egg Harbor, New Jersey
  - The Rothman Institute, Philadelphia, Pennsylvania
- Royal Blackburn Hospital, Blackburn, Lancashire, United Kingdom